CLINICAL TRIAL: NCT07342361
Title: Using Bendable Tip-suction Ureteral Access Sheath Compared to Conventional Sheath in Managing Renal Staghorn Stones A Randomized Prospective Study
Brief Title: Using Retrograde Intrarenal Surgery for Managing Staghorn Renal Stones.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Ahmed Hassan Elsergany, Principal Investigator, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 129-2025
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Renal Calculi
Keywords: staghorn calculi; retrograde intrarenal surgery; Ureteral access sheath; Suction
MeSH Terms: conditions — Kidney Calculi; Staghorn Calculi

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (1): Retrograde intrarenal surgery using a bendable tip-suction ureteral access sheath (Active Comparator): During retrograde intrarenal surgery, an ureteral access sheath with bendable tip & connected to suction system will be used.
  Interventions: Procedure: Retrograde intrarenal surgery
- Group (2): Retrograde intrarenal surgery using a conventional ureteral access sheath (Placebo Comparator): During retrograde intrarenal surgery, a conventional ureteral access sheath will be used.
  Interventions: Procedure: Retrograde intrarenal surgery

INTERVENTIONS:
Procedure: Retrograde intrarenal surgery — Retrograde intrarenal surgery with using laser for management of renal staghorn stones

SUMMARY:
This prospective, randomized study is comparing the safety and efficacy of using two types of ureteral access sheaths in managing staghorn renal stones by retrograde intrarenal surgery.

DETAILED DESCRIPTION:
Staghorn renal calculi is a complex type of renal calculi characterized by their filling of the renal pelvis and branching into all or part of the renal calyces.

Percutaneous nephrolithotomy (PCNL) is currently the recommended primary treatment option for staghorn renal calculi. However, the procedure has significant drawbacks, including invasiveness, postoperative bleeding, infection, prolonged hospitalization, and slow recovery. Retrograde Intrarenal Surgery (RIRS), an effective minimally invasive procedure, has become the first-line treatment for stones smaller than 2cm. With advancements in endoscopic equipment and techniques, RIRS is also being gradually utilized for the treatment of staghorn renal calculi in patients who are not suitable for PCNL.

Ureteral access sheath (UAS) is an important tool for the endourologist. Advantages of using a UAS in ureteroscopy include: ena¬bling repeated passage of the ureteroscope while mini¬mizing damage, improving the flow of irrigation fluid and visualization within the ureter, reducing operative times, reducing the costs of procedures and improving the effectiveness of surgery.

Intending to overcome the shortages of RIRS, a patented ureter access sheath with features of suction and bendable-tip is designed. The tip of the innovated ureteral access sheath can reach the target calyx along with the flexible ureteroscope.

The adjustable continuous negative pressure suction ensures sufficient irrigation speed and maintains a clear surgical field of view, while effectively removing fragmented stones and dust, and reducing the thermal energy generated by laser lithotripsy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes.
* Patient has a staghorn renal stone (complete or partial staghorn).
* Normal renal function tests.
* Congenital renal anomalies as horseshoe, pelvic or mal-rotated kidneys.

Exclusion Criteria:

* Abnormal coagulation profile.
* Active or untreated urinary tract infection.
* Age under 18 years or above 70 years.
* Patient has a staghorn stone associated with other pathology which requires additional intervention, as ureteral stricture or ureteropelvic junction obstruction (UPJO).
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the surgical technique | During surgery to one month after surgery
  Evaluating and comparing the incidence of operative and postoperative complications

SECONDARY OUTCOMES:
The efficacy of the surgery | One month after surgery
  Stone-free rates of the patients will be evaluated by computed tomography after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Elsergany, MSc, Principal Investigator — Helwan University
Locations (1):
- Faculty of medicine, Helwan University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bai Y, Wang X, Yang Y, Han P, Wang J. Percutaneous nephrolithotomy versus retrograde intrarenal surgery for the treatment of kidney stones up to 2 cm in patients with solitary kidney: a single centre experience. BMC Urol. 2017 Jan 18;17(1):9. doi: 10.1186/s12894-017-0200-z. PMID 28100225
- [Background] Liang H, Liang L, Lin Y, Yu Y, Xu X, Liang Z, Sheng J, Shen B. Application of tip-bendable ureteral access sheath in flexible ureteroscopic lithotripsy: an initial experience of 224 cases. BMC Urol. 2023 Nov 1;23(1):175. doi: 10.1186/s12894-023-01347-x. PMID 37915008
- [Background] Kaplan AG, Lipkin ME, Scales CD Jr, Preminger GM. Use of ureteral access sheaths in ureteroscopy. Nat Rev Urol. 2016 Mar;13(3):135-40. doi: 10.1038/nrurol.2015.271. Epub 2015 Nov 24. PMID 26597613
- [Background] Zeng G, Zhao Z, Mazzon G, Pearle M, Choong S, Skolarikos A, Denstedt J, Seitz C, Olvera Pasada D, Fiori C, Bosio A, Papatsoris A, Mendez Probst CE, Perez Fentes D, Ann Git K, Wu Q, Wiseman O, Emiliani E, Farahat Y, Ilker Gokce M, Giannakopoulos S, Goumas Kartalas I, Somani B, Knoll T, de la Rosette J, Zhong J, Vinicius Maroccolo M, Saltirov L, Chew B, Wang K, Lahme S, Giusti G, Ferretti S, Yong Cho S, Geavlete P, Cansino R, Kamphuis GM, Smith D, Matlaga BR, Ghani KD, Bernardo N, Silva AD, Ng ACF, Yang S, Gao X, Traxer O, Miernik A, Liatsikos E, Priyakant Parikh K, Duvdevani M, Celia A, Yasui T, Aquino A, Alomar M, Choonhaklai V, Erkurt B, Glass J, Sriprasad S, Osther PJ, Keeley FX Jr, Preminger GM, Cepeda Delgado M, Beltran Suarez E, Ye Z, Sarica K. European Association of Urology Section of Urolithiasis and International Alliance of Urolithiasis Joint Consensus on Retrograde Intrarenal Surgery for the Management of Renal Stones. Eur Urol Focus. 2022 Sep;8(5):1461-1468. doi: 10.1016/j.euf.2021.10.011. Epub 2021 Nov 24. PMID 34836838
- [Background] Keller EX, De Coninck V, Doizi S, Traxer O. The role of ureteroscopy for treatment of staghorn calculi: A systematic review. Asian J Urol. 2020 Apr;7(2):110-115. doi: 10.1016/j.ajur.2019.10.012. Epub 2019 Dec 5. PMID 32257803